CLINICAL TRIAL: NCT03868449
Title: Does Giving a Question Prompt List to Patients With Common Hand Conditions Improve Their Perceived Involvement in Care? A Randomized Controlled Trial
Brief Title: Question Prompt List for Common Hand Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 49833
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Carpal Tunnel Syndrome; Trigger Finger; Trigger Thumb; Dupuytren Contracture; Ganglion Cysts
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder; Dupuytren Contracture; Ganglion Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Question Prompt List (Experimental): Participants will be given a Question Prompt list that has been developed by the research team
  Interventions: Other: Question Prompt List
- 3 questions list (Active Comparator): Participants will be given 3 questions from the AskShareKnow method
  Interventions: Other: 3 questions

INTERVENTIONS:
Other: Question Prompt List — Question prompt list
  Arms: Question Prompt List
Other: 3 questions — 3 questions from the AskShareKnow model
  Arms: 3 questions list

SUMMARY:
Patients with common hand conditions will be randomized to one of two groups- one will receive a question prompt list, the other will receive a list of 3 questions

ELIGIBILITY:
Inclusion Criteria:

* patients with common hand conditions

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Perceived Involvement in Care scale | Immediately after visit
  This scale measures perceived involvement in care, with higher scores indicating higher perceived involvement

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data at this time